CLINICAL TRIAL: NCT01451905
Title: GLP-1 Receptors in Normal Skin and Skin From Patients With Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Annesofie Faurschou, MD PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLP1-PSO
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Reduction of Psoriasis Following Liraglutide Therapy in Terms of PASI and DLQI
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Psoriasis (Active Comparator)
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Victoza® is supplied in pens for injection containing 18 mg of the GLP-1 agonist liraglutide in 3 mL sterile water with disodiumphosphate and propylene glycol, and phenol for conservation (pH 8.15). Commercial pens will be used and the information given in the packaging will be applicable. The initial daily dose will be 0.6 mg for one week, 1.2 mg the following week and then 1.8 mg for the remaining treatment period. The injection is administered once daily in the morning. The maximal plasma concentration is reached 8-12 hours after subcutaneous injection. The half-life in plasma is approximately 13 hours. The duration of effect is 24 hours.
  Arms: Psoriasis
Drug: Placebo — The placebo pens contain saline and are administered in the same way and volume as Victoza. The placebo pens are specially prepared for this study and will be used in the study only
  Arms: Placebo

SUMMARY:
To examine GLP-1 receptors in skin of psoriasis patients compared with the skin of humans with no skin disease

ELIGIBILITY:
4.3 Inclusion Criteria

* Caucasians above 18 years of age
* Plaque psoriasis
* PASI score >10
* No treatment or stable treatment of psoriasis during at least 3 months before inclusion
* Steady weight through 3 months with a body mass index (BMI) above 27 kg/m2
* Normal blood pressure
* Spiral or hormonal birth control for fertile women during the entire treatment period and at least 3 days after the end of the treatment period (~5 times the plasma half-life) 4.4 Exclusion Criteria
* Psoriasis arthritis
* Fasting plasma glucose > 7.5 mmol/L or HbA1c > 7.5%
* Type 1 diabetes
* Treatment for type 2 diabetes with GLP-1-based medicine (DDP-4-inhibitors or GLP-1-receptor-agonists)
* Heart failure, NYHA class III-IV
* Uraemia, end-stage renal disease, or any other cause of impaired renal function with s-creatinine >150 µM and/or albuminuria
* Liver disease (alanine amino transferase (ALAT) and/or aspartate amino transferase (ASAT) >2 x upper normal serum levels)
* Anaemia
* Acute or chronic pancreatitis
* Struma or thyroid cancer
* Pregnancy or breast feeding
* Inability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Changes in PASI and DLQI | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark